CLINICAL TRIAL: NCT00747656
Title: The Impact of Prehospital 12 Lead ECG With Advanced Emergency Department Notification on Time to In-hospital Reperfusion Strategy in Patients With Acute ST Segment Elevation Myocardial Infarction - A Prospective Study
Brief Title: Prehospital Evaluation and Economic Analysis of Different Coronary Syndrome Treatment Strategies - PREDICT
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Daria O'Reilly, Associate Professor, St. Joseph's Healthcare Hamilton
Other Study IDs: HTA006-0708-01
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Myocardial Ischemia; Myocardial Infarction
Keywords: Electrocardiography; Emergency medical services; Emergency medicine; Health services; Cost effectiveness
MeSH Terms: conditions — Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: 3 lead ECG subjects with chest pain and suspected ischemia transported to the nearest receiving ED and not eligible for bypass based on transport time
- 2: 3 lead ECG subjects with chest pain and suspected ischemia transported to the nearest receiving ED and eligible for bypass based on transport time, if 12 lead PHECG was possible
- 3: 12 lead ECG subjects with prehospital notification transported to nearest receiving ED adn not eligible for bypass to PCI center based on transport time
- 4: 12 lead PHECG subjects with prehospital notification bypassed past the nearest receiving ED to the PCI center.

SUMMARY:
Despite remarkable gains in treatment over the last decade short-term mortality for those who survive to hospital with AT-elevation acute myocardial infarction (STEMI) remains high (5%-10%). Different studies have pointed out that reperfusion (intravenous fibrinolysis or percutaneous coronary interventions (PCI) and its timing are critical in decreasing STEMI patients' mortality. Studies of prehospital 12 lead electrocardiograms (12 lead PHECG) with advance emergency department (ED) notification suggest that there is a time to treatment advantage with this intervention. The use of 12 lead PHECG is not currently universal and part of standard treatment throughout the province. The purpose of the study is to follow STEMI study subjects during standard treatments and to compare the outcomes of subjects that received 12 lead PHECG with advanced ED notification in mixed rural/urban areas with outcomes of subjects treated in areas with only 3 lead PHECG monitoring and indirect ED notification. The investigators hypothesize that there will be a survival benefit for study subjects with 12 lead PHECG and advance ED notification in rural and urban environments through a reduction in door-to-reperfusion time and that 12 lead PHECG will be a cost-saving technology for the province of Ontario.

DETAILED DESCRIPTION:
Many studies have established that reperfusion reduces mortality in ST-elevation acute myocardial infarction (STEMI) patients; the earlier reperfusion therapy is delivered, the greater the mortality reduction. Most STEMI patient in Ontario still do not receive reperfusion therapy within established target times of <30 minutes for fibrinolysis or <90 minutes for PCI. 12 lead PHECG with advance ED notification may have a time to treatment impact in STEMI patients. However studies, investigating this intervention were all small, largely urban trials, and were carried out with advanced care paramedics. In Ontario, many emergency medical services (EMS) systems cover large rural regions, and are frequently staffed by primary care paramedics with only basic life support training. Thus, the benefit of 12 lead PHECG in these settings is unclear. In addition, no study has assessed the cost-effectiveness of 12 lead PHECG compared to 3 lead PHECG.

ELIGIBILITY:
Inclusion Criteria:

* Call 911 for assistance
* Are suspected by the paramedics of having ischemic chest pain for greater than 30 minutes but less than 6 hours
* Be greater than or equal to 18 years of age
* Experience chest pain that fails to completely respond to nitrates as per standard provincial chest pain protocol.

Exclusion Criteria:

* Subjects less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted across Ontario. Selected regions representing approximately 17% of the population of Ontario and 6.4% of the popluation of Canada. Covering an area of 181426 per square kilometers with variable population densities from 2.5 to 234 person per square kilometers and representing rural, suburban, urban, and metropolis areas will be the catchment area for the study. A variety of EMS operators under the control of EMS Base Hospital programs will be involved in the data collection for this study. Patients presenting with suspected ischemic chest pain will be tracked as a part of the trial.
Sampling Method: Non-Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2009-02; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the time from arrival to the ED to initiation of the reperfusion therapy between those receiving 12 lead PHECG and those receiving 3 lead PHECG monitoring prior to hospital arrival. | 24 hours

SECONDARY OUTCOMES:
Survival at 30 days | 30 days
Cost-effectiveness | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Morrison, MD, MSc, Principal Investigator — Prehospital & Transport Medicine Research, Sunnybrook Health Sciences Centre; Ron Goeree, MA, Principal Investigator — Programs for Assessments of Technology in Health Reasearch Institute, St. Joseph's Healthcare Hamilton
Locations (5):
- Canada (5):
  - Stevenson Memorial Hospital, Alliston, Ontario
  - Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Rouge Valley, Toronto, Ontario
  - Sunnybrook Health Scineces Centre, Toronto, Ontario

REFERENCES:
- [Background] Morrison LJ, Rac VE, Bowen JM, Schwartz B, Perreira T, Ryan W, Zahn C, Chadha R, Craig A, O'Reilly D, Goeree R. Prehospital evaluation and economic analysis of different coronary syndrome treatment strategies--PREDICT--rationale, development and implementation. BMC Emerg Med. 2011 Mar 29;11:4. doi: 10.1186/1471-227X-11-4. PMID 21447161
- See also: Programs for Assessments of Technology in Health Research Institute — http://www.path-hta.ca/